CLINICAL TRIAL: NCT06417086
Title: Clinical Evaluation of Acupuncture Treatment on Alzheimer's Disease in APOE e4 Carriers and Non-Carriers: A Randomized Controlled Trial
Brief Title: Clinical Evaluation of Acupuncture Treatment on Alzheimer's Disease in APOE e4 Carriers and Non-Carriers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ZhanYJ (Other)
Collaborators: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor-Investigator, ZhanYJ, Shanghai University of Traditional Chinese Medicine, Shanghai University of Traditional Chinese Medicine
Organization: Shanghai University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23Y11921000
Record Dates: First submitted 2024-05-12; First posted 2024-05-16 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Acupuncture Therapy; Donepezil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Streitberger placebo needle will be used as sham acupuncture method to mask the paticipants. The outcome assessors will also be blind to the grouping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture Treatment (Experimental): Participants in this group will receive acupuncture treatment in combination with donepezil for 12 weeks.
  Interventions: Other: Acupuncture; Drug: Donepezil
- Sham Acupuncture Treatment (Active Comparator): Participants in this group will receive sham acupuncture treatment in combination with donepezil for 12 weeks.
  Interventions: Other: Sham Acupuncture; Drug: Donepezil

INTERVENTIONS:
Other: Acupuncture — The main acupoints are DU 24, EX-HN 3, DU 20, EX-HN 1, GB 12, HT 7, KI 6, GB39, and then selecting other acupoints according to TCM syndrome. There will be 12 weeks of 3-session treatment for each participant in total.
  Arms: Acupuncture Treatment
Other: Sham Acupuncture — The Streitberger placebo needle will be used to simulate an acupuncture procedure without penetrating the skin. The main acupoints are DU 24, EX-HN 3, DU 20, EX-HN 1, GB 12, HT 7, KI 6, GB39, and then selecting other acupoints according to TCM syndrome. There will be 12 weeks of 3-session treatment for each participant in total.
  Arms: Sham Acupuncture Treatment
Drug: Donepezil — Donepezil 5 mg will be given once daily before bed-time for 12 weeks.

SUMMARY:
The goal of this clinical trial is to learn if acupuncture works to treat mild-to-moderate Alzheimer's disease, as well as the difference of its effect in APOE e4 carriers and non-carriers. It will also learn about the safety of acupuncture.

Researchers will compare acupuncture to a placebo (sham acupuncture) to see if acupuncture works to relieve the cognitive impairment and improve the ability of daily living and the quality of life. In addition, the plasma and neuroimaging biomarkers will be included as objective indexes.

Participants will:

Experience acupuncture or sham acupuncture 3 times per week for 12 weeks, and receive a 52-week follow-up.

Visit the clinic at Week 12, Week 38 and Week 64 for checkups and tests.

DETAILED DESCRIPTION:
This is a two-centre randomized controlled trial. A total of 176 participants with mild-to-moderate Alzheimer's disease, 88 APOE e4 carriers and 88 non-carriers, will be randomly assigned to either an acupuncture combined with donepezil group or a sham acupuncture combined with donepezil group with a ratio of 1:1. The main acupoints are DU 24, EX-HN 3, DU 20, EX-HN 1, GB 12, HT 7, KI 6, GB39. There will be 12 weeks of 3-session treatment for each participant, and a 52-week follow-up in total. The primary outcome is the change and effective rate from baseline in the ADAS-cog score measured at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 50-85 years
* Diagnosed by the criteria of Neurological Communicative Disorders and Stroke and the Alzheimer Disease and Related Disorders Association (NINCDS-ADRDA)
* Cognitive impairment based on the scores of the Chinese version of the Mini Mental State Examination (MMSE) (patients with mild to moderate Alzheimers disease, 11≤primary school degree≤22, 11≤junior high school degree or above≤26
* Magnetic resonance imaging (MRI) confirmation of atrophy of the hippocampus or the medial temporal lobe volume, MRI manifestation of high possibility of Alzheimer Disease
* The Medial Temporal Lobe Atrophy Rating Scale (MTA-scale) score (≥2 for those under 75 years, and ≥3 for those over 75 years)
* Voluntarily joining this study with informed consents

Exclusion Criteria:

* Cognitive impairment caused by other factors (e.g. vascular dementia, dementia with Lewy bodies, frontotemporal dementia, hormone or metabolic abnormalities, hypothyroidism, folic acid or vitamin B12 deficiency, delirium or other mental and emotional disorders (such as schizophrenia and depression))
* A serious heart condition, hepatic disease, renal system disease, hematopoietic system disease, or whole-body malnutrition
* Aphasia, disturbance of consciousness, or failure to cooperate with the related examinations due to physical disability
* Contraindications to undergoing an MRI scan such as claustrophobia or pacemaker implantation.
* Anticoagulant treatments such as warfarin or heparin
* Use of pacemakers or receiving acupuncture in the past 2 weeks

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognition (ADAS-cog) | Change from baseline to Week 12
  The maximum score of the ADAS-cog is 70 including 12 items. The questions in this scale contain word recall task, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition task, remembering test directions, spoken language, word-finding difficulty, comprehension and attention. In general, a normal score for someone who does not have AD or another type of dementia is 5. The higher scores indicate higher degree of cognitive dysfunction.

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognition (ADAS-cog) | Change from baseline to Week 38 (Follow-up 1) and Week 64 (Follow-up 2)
  The maximum score of the ADAS-cog is 70 including 12 items. The questions in this scale contain word recall task, naming objects and fingers, following commands, constructional praxis, ideational praxis, orientation, word recognition task, remembering test directions, spoken language, word-finding difficulty, comprehension and attention. In general, a normal score for someone who does not have AD or another type of dementia is 5. The higher scores indicate higher degree of cognitive dysfunction.
Alzheimer's Disease Cooperative Study-Activity of Daily Living (ADCS-ADL) | Change from baseline to Week 12, Week 38 (Follow-up 1) and Week 64 (Follow-up 2)
  The maximum of the ADCS-ADL score is 54 containing 19 domains about assessment of basic and operational ability of daily living. The higher scores indicate higher ability of daily living.
Quality of Life-Alzheimer's Disease(QOL-AD) | Change from baseline to Week 12, Week 38 (Follow-up 1) and Week 64 (Follow-up 2)
  The QOL-AD score includes 13 items about physical health, mental health, social and financial assessment, and quality of life. The total score ranges from 13 to 52. The higher scores indicate higher quality of life.

OTHER OUTCOMES:
Phosphorylated tau at threonine 181 (p-tau181) | Change from baseline to Week 12 and Week 64 (Follow-up 2)
  Plasma p-tau181measured by Single Molecule Array (Simoa) as the plasma biomarker.
Cerebral Blood Flow (CBF) | Change from baseline to Week 12 and Week 64 (Follow-up 2)
  CBF acquired by arterial spin labeling (ASL) magnetic resonance imaging (MRI) technique measures the blood flow condition of the whole brain.

CONTACTS AND LOCATIONS:
Overall Officials: Yijun Zhan, Study Chair — Shanghai University of Traditional Chinese Medicine; Houguang Zhou, Study Director — Huashan Hospital
Locations (1):
- Longhua Hospital, Shanghai University of Traditional Chinese Medicine, Shanghai, China